CLINICAL TRIAL: NCT06447220
Title: Washed Microbiota Transplantation for Malnutrition
Status: Recruiting | Type: Observational
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Other Study IDs: WMT-MN-2024
Record Dates: First submitted 2024-05-19; First posted 2024-06-07 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2024-07

CONDITIONS: Malnutrition
Keywords: washed microbiota transplantation; malnutrition; fecal microbiota transplantation
MeSH Terms: conditions — Malnutrition | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — fecal, blood and urine samples before and 12 weeks after washed microbiota transplantation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- The malnourished undergoing washed microbiota transplantation: patients undergoing washed microbiota transplantation who were diagnosed as malnutrition according to weight loss or low BMI
  Interventions: Procedure: washed microbiota transplantation
- The malnourished not undergoing washed microbiota transplantation: The malnourished patients did not undergo washed microbiota transplantation

INTERVENTIONS:
Procedure: washed microbiota transplantation — The prepared microbiota suspension was infused into the patients' gut.
  Other Names: fecal microbiota transplantation
  Groups: The malnourished undergoing washed microbiota transplantation

SUMMARY:
Malnutrition is a pathological condition in which dietary intake fails to meet the body's energetic or nutritional needs. It may be caused by macronutrient or micronutrient deficiencies, high energy expenditure, impaired nutrient absorption or assimilation. Malnutrition can affect all stages of life. In adults, malnutrition is strongly associated with poor clinical outcomes such as increased morbidity, increased mortality and prolonged hospitalization. In children, malnutrition can lead to growth retardation, cognitive impairment and immune dysfunction.

DETAILED DESCRIPTION:
The gut microbiota of malnourished patients is different from that of healthy people. The diversity of the gut microbiota of patients with severe malnutrition reduced and the abundance of Proteobacteria significantly increased, as well as pathogenic genera such as Klebsiella, Escherichia coli, Shigella, and Streptococcus. This suggests that gut microbiota plays an important role in the occurrence and development of malnutrition. Dietary intervention targeting gut microbiota can quickly improve children's malnutrition, promote weight gain and increase protein levels that promote bone growth and nerve development. Exclusive enteral nutrition combined with immediate washed microbiota transplantation(WMT) can rapidly improve the nutritional status of patients with Crohn's disease compared with those with delayed WMT. Gut microbiota has been confirmed to be closely related to malnutrition. Improving the disordered gut microbiota in malnourished patients may become a potential treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Meet any of the following two conditions: ①weight loss (>5% weight loss in the past 6 months or >10% weight loss in more than 6 months); ②low BMI (<70 years old and BMI<18.5kg/m2 or ≥70 years old and BMI<22kg/m2);
3. Underwent washed microbiota transplantation.

Exclusion Criteria:

1. Expected survival time <3 months;
2. Women who are pregnant or breastfeeding;
3. Other patients deemed not suitable for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malnutrition receiving WMT will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-17 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
change of the third lumbar vertebrae skeletal muscle mass and height | baseline, 12 weeks post transplantation
  The third lumbar vertebrae skeletal muscle mass represents the sum of the cross-sectional areas of the skeletal muscles at the L3 level, including the psoas major, the erector spinae, the quadratus lumborum, the musculus transversus abdominis, the obliquus externus abdominis and the obliquus internus abdominis. Skeletal muscle mass and height will be combined to report the third lumbar vertebrae skeletal muscle mass index(L3 SMI) in cm^2/m^2.
change of weight and height | baseline, 4 weeks, 8 weeks, 12 weeks post transplantation
  Weight and height will be combined to report BMI in kg/m^2.

SECONDARY OUTCOMES:
change of the 5-level EuroQoL Group's 5-dimension (EQ-5D-5L) | baseline, 4 weeks, 8 weeks, 12 weeks post transplantation
  EQ-5D-5L is a 5-dimension questionnaire measuring health state and each dimension represents the level from 1 to 5, with higher level indicating worse health state.
change of the Pittsburgh Sleep Quality Index (PSQI) | baseline, 4 weeks, 8 weeks, 12 weeks post transplantation
  PSQI is a self-rated questionnaire which assesses sleep quality over a 1-month time interval. Nineteen items generate seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for seven components yields one global score, with higher score indicating worse sleep quality.
change of the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) | baseline, 4 weeks, 8 weeks, 12 weeks post transplantation
  FACIT-Fatigue is a 13-item test measuring fatigue and each item receives a value from 0 to 4, with higher value indicating worse fatigue state.
change of the Gastrointestinal Symptom Rating Scale(GSRS) | baseline, 4 weeks, 8 weeks, 12 weeks post transplantation
  GSRS is a 13-item test to make a comprehensive assessment of common gastrointestinal symptom and each item receives a value from 0 to 3, with higher value indicating worse gastrointestinal condition.
change of insulin-like growth factor I(IGF-I) | baseline, 12 weeks post transplantation
  Blood is tested for Insulin-like growth factor I.
the difference of the gut microbiota composition before and after washed microbiota transplantation | baseline, 12 weeks post transplantation
  The composition of the gut microbiota is evaluated by sequencing faecal metagenome. We evaluate the differences in the structure of the flora and its metabolism.
the incidence of treatment-related adverse events (AE) assessed by CTCAE, Version 5.0 | 12 weeks post transplantation
  The severity of AE was graded as mild (grade 1), moderate (grade 2), severe/disabling (grade 3), life threatening (grade 4), and death (grade 5). All AE were divided in definitely, probably and possibly related to treatment. The treatment-related AE we focused on included microbiota-related AEs (e.g., infection, diarrhea, abdominal pain, etc.) and route of delivery related AEs (e.g., nausea, vomiting, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Department of Microbiota Medicine & Medical Centre for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller J, Wells L, Nwulu U, Currow D, Johnson MJ, Skipworth RJE. Validated screening tools for the assessment of cachexia, sarcopenia, and malnutrition: a systematic review. Am J Clin Nutr. 2018 Dec 1;108(6):1196-1208. doi: 10.1093/ajcn/nqy244. PMID 30541096
- [Background] Dent E, Wright ORL, Woo J, Hoogendijk EO. Malnutrition in older adults. Lancet. 2023 Mar 18;401(10380):951-966. doi: 10.1016/S0140-6736(22)02612-5. Epub 2023 Jan 27. PMID 36716756
- [Background] Fontaine F, Turjeman S, Callens K, Koren O. The intersection of undernutrition, microbiome, and child development in the first years of life. Nat Commun. 2023 Jun 15;14(1):3554. doi: 10.1038/s41467-023-39285-9. PMID 37322020
- [Background] Coley EJL, Hsiao EY. Malnutrition and the microbiome as modifiers of early neurodevelopment. Trends Neurosci. 2021 Sep;44(9):753-764. doi: 10.1016/j.tins.2021.06.004. Epub 2021 Jul 21. PMID 34303552
- [Background] Chen RY, Mostafa I, Hibberd MC, Das S, Mahfuz M, Naila NN, Islam MM, Huq S, Alam MA, Zaman MU, Raman AS, Webber D, Zhou C, Sundaresan V, Ahsan K, Meier MF, Barratt MJ, Ahmed T, Gordon JI. A Microbiota-Directed Food Intervention for Undernourished Children. N Engl J Med. 2021 Apr 22;384(16):1517-1528. doi: 10.1056/NEJMoa2023294. Epub 2021 Apr 7. PMID 33826814
- [Background] Xiang L, Yu Y, Ding X, Zhang H, Wen Q, Cui B, Zhang F. Exclusive Enteral Nutrition Plus Immediate vs. Delayed Washed Microbiota Transplantation in Crohn's Disease With Malnutrition: A Randomized Pilot Study. Front Med (Lausanne). 2021 Oct 22;8:666062. doi: 10.3389/fmed.2021.666062. eCollection 2021. PMID 34746161